CLINICAL TRIAL: NCT07197190
Title: Hybrid Autologous Breast Augmentation in Mastopexy With Internal BRA Fixation; Using Local Breast Tissues and Fat Grafting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Hassan M. Elhawary, Plastic surgery Specialist, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Augmentation mastopexy
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Ptosis
Keywords: Internal Bra; Sub-pectoral lipofilling; Autologous Augmentation mastpexy; Breast fat grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female patient with breast ptosis, grade 2 or 3, with small or medium sized breast. (Experimental): - Study subjects:
  1. Inclusion criteria:
     1. Female patient
     2. Grade 2 or 3 breast ptosis according to Regnault classification.
     3. Age is between 18 years and 50 years old.
     4. Small to moderate breast size.
  2. Exclusion criteria:
     1. Age is below 18 years and above 50 years.
     2. Pregnant or breast-feeding patient.
     3. Large sized breast.
     4. Grade 1 breast ptosis or pseudoptosis according to Regnault classification.
     5. Patients are currently under treatment of breast cancer.
     6. Immunosuppressed patients. They are all subjected to autologous augmentation mastopexy with subpectoral lipofilling and upper and medial pole fat grafting.
  Interventions: Procedure: Autologous augmentation mastopexy with subpectoral lipofilling and upper and medial pole fat grafting.

INTERVENTIONS:
Procedure: Autologous augmentation mastopexy with subpectoral lipofilling and upper and medial pole fat grafting. — The term 'internal bra' refers to a range of techniques that aim to stabilise the position of the breast and improve longevity of surgical results. In this study, the investigators address one of them which is dermal flap technique. Dermal flaps have two key advantages, the first of which is that they are low cost due to their autologous nature. The fact that they utilise the patient's own tissue also means they are not associated with an increased risk of infection or immunological reaction, which is their second main advantage, But it has some drawbacks on the long term, such as upper pole hollowness and lack of breast parenchymal tissue to give a good breast volume.
  In this research, the investigators used the autogenous internal BRA mastopexy technique for correction of breast ptosis and sub pectoral lipofilling to help increase the breast volume and subcutaneous fat grafting to give the breast upper pole fullness.

SUMMARY:
The breast is a very important organ for women's self-esteem and is regarded as a symbol of femininity. Deviations from normal size, shape, and symmetry are interpreted as unattractive and a sign of aging. Far from posing merely a cosmetic problem, such deviations deeply disturb both the patient's perception of her body and her emotional balance.

The first breast surgeries started as early as the 6th century, yet the aesthetic breast surgeries and specifically mastopexy techniques were first recorded in the 19th century in parallel with the evolution of reduction mammaplasty. Most of these techniques involved suspension targeting breast mound elevation.

Breast ptosis refers to the downward displacement of the nipple-areola complex (NAC) below the inframammary fold (IMF), commonly due to aging, pregnancy, weight fluctuations, and genetics. It's caused by loss of skin elasticity, stretching of Cooper's ligaments, parenchymal involution, and genetic factors. The degree of ptosis can be categorized by the Regnault classification, which assesses the breast according to the relative position of the nipple to the inframammary fold (IMF):

Grade 1: Mild ptosis - The nipple is at the level of the IMF. Grade 2: Moderate ptosis - The nipple is below the level of the IMF but is not the most dependent part of the breast.

Grade 3: Severe ptosis - The nipple is below the IMF and is the most dependent part of the breast.

Pseudoptosis designates a breast configuration in which the nipple is located above or at the level of the IMF, most of the breast is well below the IMF, and the nipple-to-IMF distance is often greater than 6 cm.

Mastopexy procedures are similar and traditionally derived from reduction procedures, involving skin resection with no or minimal parenchymal resection. There are three main surgical goals that should be attained to correct breast ptosis and give a firm aesthetic breast shape. These include nipple areola complex (NAC) elevation, skin envelope excess management and breast reshaping. Breast flaps and parenchymal shaping manoeuvres can help auto augmentation correct any shape defects, Hence come the idea of autogenous internal bra mastopexy technique.

The term 'internal bra' refers to a range of techniques that aim to stabilise the position of the breast and improve longevity of surgical results. They can be categorised into 5 groups: mesh techniques, acellular dermal matrix (ADMs) techniques, suture techniques, dermal flap techniques, and muscle techniques. In this study, the investigators address one of the dermal flap techniques. Dermal flaps have two key advantages compared to meshes and ADMs, the first of which is that they are low cost due to their autologous nature The fact that they utilise the patient's own tissue also means they are not associated with an increased risk of infection or immunological reaction, which is their second main advantage.

There are many different types of pedicled flaps in mastopexy as medial, superior and superomedial flaps. But in this study, the investigators use the superior pedicelled flap with inferior dermal flap described by Liacyr Ribeiro.

This flap can be better mobilized than any of the other flaps, and the breast and the flap move together. The flap does not heal to pectoralis fascia; rather, the anterior surface of the flap heals to the posterior surface of the pedicle. Later, if the patient decides to have an implant, there is still a good plane between the pectoralis fascia and the inferior flap. This plane could be filled by sub pectoral fascia fat grafting.

Autologous augmentation mastopexy may seem the most suitable technique for ptotic small sized breasts. But it has some drawbacks on the long term, such as upper pole hollowness. This issue can also be addressed by upper pole fullness by fat grafting.

So, in this research, the investigators do autologous internal bra mastopexy with fat grafting in two planes: Sub- fascial level for augmentation and subcutaneous level for upper pole fullness. The investigators assess the result by taking pre and post operative breast measurements and photographs. The investigators also assess participants' satisfaction level and possible complication.

DETAILED DESCRIPTION:
*Aim of work: To achieve breast autologous internal BRA mastopexy in grade 2 and 3 breast ptosis using, auto-augmentation with tissue rearrangement, sub pectoral fascia fat grafting and upper pole lipofilling. And 6-month long follow-up to observe participants' satisfaction level, measurements and complications.

*Patients and Methods: A primary prospective randomized control trial. Inclusion criteria

1- Female patient. 2- Grade 2 or 3 breast ptosis according to Regnault classification. 3- Age is between 18 years and 50 years old. 4- Small and medium sized breast. Exclusion criteria

1. Age is below 18 years and above 50 years.
2. Pregnant or breast-feeding patient.
3. Large sized breast.
4. Grade 1 breast ptosis or pseudoptosis according to Regnault classification.
5. Patients are currenting under treatment of breast cancer.

   * Patient Sheet

     1. Pre-operative data:

        Personal History: Name, age, sex, Job, Marital status, co-morbidities and smoking.

        Preoperative investigations: blood count, coagulation profile, basic metabolic panel and mammograms.
     2. Examination:

        - It included body mass index, abdominal examination (site of liposuction for fat grafting) and breast examination.
        * Breast measurements while standing in a lateral position include

<!-- -->

1. Suprasternal notch to nipple (SN-N)
2. Inframammary fold distance.
3. Base width
4. Areola diameter
5. Inter-nipple distance.
6. nipple to inframammary fold (N-IMF).
7. Upper pole projection.
8. Lateral maximum projection.
9. Humerus length. Finally, circumference measurements were obtained at three different levels: upper pole, level of maximum projection and at the level of IMF.

   - Preoperative photographs were taken for each patient in anterior, oblique and lateral views. 2*Operative data: Markings
   * The preoperative drawings proceed with the patient in standing position.
   * The surgical procedure is done using an inverted-T approach preserving a superior pedicle for the blood supply of the nipple-areola complex (NAC).

<!-- -->

1. The sternal notch with the mid sternal line, the inframammary crease line and the mid breast line.
2. The new nipple position is located on the mid breast line at the level of the inframammary fold on the anterior surface of the breast.
3. The mid breast line is marked from the clavicle to the nipple and then continued from the inframammary crease down the lower thoracic wall.
4. Then, by moving the breast gently with the hand medially and laterally the new position of the nipple is connected by drawing a vertical line to the mid breast line at the level of the inframammary fold marking. The more the breast is moved either laterally or medially, the wider the angle of the inverted V becomes, this is directly correlated with the amount of resected skin.
5. On both lines of the inverted V drawing two marks are set on each line, the first about 5cm from the new NAC position, and the second one another 6cm away from the first mark. The first marks relate to each other using a semicircular line that is drawn 1.5cm above the new nipple position on the mid breast line. This point is the new apex of the NAC. The secondary marks are connected horizontally with the inframammary crease line medially and laterally.
6. Within this marking the superior pedicle is designed starting from the new NAC apex. The base of the superior pedicle should not measure less than 8cm. The symmetry of the markings, especially the new NAC positions, are checked in front of a mirror.

Surgical procedure:

- The patient is put under general anesthesia in supine position.

- After marking the incisions and new nipple position, the areola was slightly stretched and marked with a 5 cm cookie cutter.

- The peri areolar area to new nipple position and wedge-shaped vertical segments were deepithelialized for preparation of the flap for auto augmentation.

* The superior curved border of the lower island flap is cut from the lower aspect of the areola. Dissection using diathermy is done vertically downwards till pectoralis major fascia was seen. while the breast was held by the surgical assistant keeping it in place and not falling laterally.
* During dissection of the superior border, two wings corresponding to curvature of areola were kept as part of the flap. The lateral vertical border of the flap was dissected subcutaneously till anterior axillary line to help decrease the lateral fullness of the breast.
* The medial border, however, was divided vertically downwards to the pectoralis fascia, leaving the medial fullness of the breast intact. As with the superior border, dissection was done with the breast supported by a surgical assistant
* The inferior flap was partially separated by cutting the dermal end of the flap. A sub glandular pocket was then directed upwards and medially reaching the marked superior border of the breast, with a width equal to superior border flap length.
* After hemostasis, Sub fascial fat grafting is done of previously harvested adipose tissue, using size 2 and 3 mm canula with 50 cc interlocked syringe.

Then the flap was transposed superiorly, and three separate sutures were taken between upper borders of flap and pectoralis muscle and fascia using polypropylene 1 or zero.

* The NAC was attached at the 12 o'clock point at the new nipple position and the vertical lines were approximated together. The stapled vertical line was pulled and stretched, showing the excess skin envelope, which was marked and excised.
* The new NAC is marked using a cookie cutter at the most projecting point of the lifted breast.
* Skin is closed using Vicryl 2-0 and 3-0 for subcutaneous tissue and Vicryl 4-0 for dermis.
* After subcutaneous tissue closure, the upper pole is evaluated and the 2nd fat injection is done, in a fanning mode in subcutaneous level.
* No drains are needed.
* Dressing is done by Steri- strip in a vertical pattern, then a soft bra is used.

Liposuction and fat harvesting procedure:

- The donor areas for lipo-aspiration are mainly lower abdomen and thighs. The patient's choice is taken into consideration.

* Infiltration of the area is done using Tumescent technique:

For each 500 cc of Ringer solution, the investigators add 1 mL of epinephrine and 10 cc of 2% Lidocaine.

* Aspiration was done using a wide bore 4 mm cannula.
* Fat was processed by sedimentation.
* After about 20 minutes adipose portion of separated fat is transferred to 20-ml syringes.

  3*Postoperative Care
* A change of dressing is carried out after 24 hours.
* Skin stitches are usually absorbed within 3 weeks. Postoperatively.
* Patients were instructed to lie supine and refrain from using the breast for a period of at least three months.

  4*Post-operative data:
  1. Breast measurements: the same measurements that were taken preoperatively.
  2. patient satisfaction level: which is measured using a Breast Q questionnaire.
  3. Photographic Documentation: At the same positions taken preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient
2. Grade 2 or 3 breast ptosis according to Regnault classification.
3. Age is between 18 years and 50 years old.
4. Small to moderate breast size.

Exclusion Criteria:

1. Age is below 18 years and above 50 years.
2. Pregnant or breast-feeding patient.
3. Large sized breast.
4. Grade 1 breast ptosis or pseudoptosis according to Regnault classification.
5. Patients are currently under treatment of breast cancer.
6. Immunosuppressed patients. -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Photpgraphs | Preoperative, postoperative and 6- month follow-up.
  Photographs were taken for each patient in anterior, oblique and lateral views.
Breast measurements. | Pre- operative, post operative and 6- month follow up.
  Breast measurements while standing in a lateral position include
  1. Suprasternal notch to nipple (SN-N)
  2. Inframammary fold distance.
  3. Base width
  4. Areola diameter
  5. Inter-nipple distance.
  6. nipple to inframammary fold (N-IMF).
  7. Upper pole projection.
  8. Lateral maximum projection.
  9. Humerus length. Finally, circumference measurements were obtained at three different levels: upper pole, level of maximum projection and at the level of IMF.
Patient statisification level | Pre-operative, postoperative and after 6 month.
  Patient statisification level is measured using a breast q questionaire. The improvement postoperative is measured by increased statisification and quality of life than preoperative assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut unversity Hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
For patients' privacy.

REFERENCES:
- See also: Breast Q test, the measurement tool for patients' statisfication. — https://patientreportedoutcomes2.sites.olt.ubc.ca/files/2014/04/BREAST-Q-ReductionMastopexyModule-Postoperative_AU1.0_eng-USori.pdf